CLINICAL TRIAL: NCT00361738
Title: A Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, Dose-Response, Multicentre, Multinational Study Evaluating the Efficacy and Safety of AVE2268 Administered Either Twice Daily (Breakfast and Lunch) at a Dose of 300, 600 and 1200 mg or Once Daily (Breakfast) at a Dose of 1200 mg, in Patients With Type 2 Diabetes Treated With Metformin and Not Adequately Controlled
Brief Title: Dose-Ranging Study Evaluating AVE2268 in Patients With Type 2 Diabetes Not Adequately Controlled by a Metformin Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DRI6738; EUDRACT: 2006-001843-74
Record Dates: First submitted 2006-08-07; First posted 2006-08-08 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2009-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — AVE2268

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: AVE2268

SUMMARY:
Dose-ranging study of AVE2268 in the management of patients with type 2 diabetes mellitus also receiving metformin.

Its main objectives will be to assess the effects of several doses of AVE2268 on Mean Plasma Glucose. Its secondary objectives will be to assess the effects of AVE2268 on plasma glucose (fasting and post-prandial), and also the safety and tolerability of AVE2268.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus, as defined by the American Diabetes Association, for at least one year at the time of screening.
* HbA1c measured at visit 1 in the range of ≥ 7.0 and < 9.0 %.
* Stable metformin treatment (dose ≥ 1.5g/day for at least 3 months prior to enrollment in the study). No other antidiabetic medications are permitted for 3 months prior to enrollment.

Exclusion Criteria:

* Pregnant or breast-feeding women.
* Women of childbearing potential not protected by medically approved contraceptive method of birth control.
* BMI >40kg/m2
* Diabetes other than type 2 diabetes.
* Subjects with "brittle-diabetes" or any hospitalization or emergency room visit due to poor diabetic control within the past 6 months, previous history of diabetes related dehydration leading to hospitalization, history or evidence of ketoacidosis.
* Presence or history of cancer within the past five years.
* Evidence within the past 6 months of myocardial infarction, stroke, retinopathy requiring laser surgery, or heart failure requiring hospitalization.
* Impaired hepatic tests, impaired renal function.
* History or evidence of clinically relevant renal or urological disorder.
* The investigator will evaluate whether there are other reasons why a patient may not participate.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2006-07; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Change in Mean Plasma Glucose (MPG) from baseline to week 4.

SECONDARY OUTCOMES:
Glucose parameters (change from baseline to week 4 in fasting and post prandial plasma glucose) ; Change in HbA1c and fructosamine ; Safety: physical examination, adverse events, ECG, laboratory tests

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth SOUHAMI, M.D, Study Director — Sanofi
Locations (11):
- Sanofi-Aventis Administrative Office, San Isidro, Argentina
- Sanofi-Aventis Administrative Office, Cove, New South Wales, Australia
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, Hørsholm, Denmark
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Midrand, South Africa

REFERENCES:
- See also: Related Info — http://www.sanofi-aventis.com